CLINICAL TRIAL: NCT00712153
Title: Follow-up of Coronary Artery Bypass Graft Patency by Multislice Computed Tomography
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shih-Hong Huang, Far Eastern Memorial Hospital
Other Study IDs: 95023; FEMH - 95 - D -001
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease
Keywords: multislice computed tomography; coronary artery bypass grafting; Patients; underwent; surgeries
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary artery disease is a major cause of morbidity and mortality across the world and coronary artery bypass surgery (CABG) is the most common surgical procedure for treatment. Patients with recurrent ischemic symptoms after CABG are most likely to have occluded or significantly stenosis in grafts or native coronary arteries. Therefore, there is a need to evaluate the patency of these vessel conduits after CABG. Until now, selective coronary angiography is the traditional gold standard for the assessment of both native coronary arteries and bypass grafts. But it is an invasive procedure that requires x-ray exposure, hospitalization, and includes a risk for complication. However, there is an alternative noninvasive method, multislice computed tomography (MSCT), with high specificity and excellent sensitivity for the detection of the coronary artery disease. It is even cheaper and takes shorter time to perform. Accordingly, the purpose of this study is to use MSCT to evaluate the patency and the quality of all grafts and native coronary arteries after CABG for more than two years. In addition, we will elucidate the relationship of these data and CABG procedures to review our experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent CABG and performed MSCT after the surgeries

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent CABG and performed MSCT after the surgeries
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual)